CLINICAL TRIAL: NCT03439930
Title: The Effect of Balance Training on Neuromuscular Control in Subjects With CAI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015/0711
Record Dates: First submitted 2018-02-14; First posted 2018-02-20 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Ankle Inversion Sprain; Instability, Joint; Treatment; Neuromuscular Control; Reaction Time
MeSH Terms: conditions — Joint Instability

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Uni-axial (Active Comparator): Subjects in this group perform exercises on an uni-axial balance board
  Interventions: Other: Balance training
- Multidirectional (Active Comparator): Subjects in this group perform exercises on a multidirectional balance board
  Interventions: Other: Balance training

INTERVENTIONS:
Other: Balance training — 6 weeks lasting balance training program

SUMMARY:
The goal of this study is evaluate the effect of uni-axial versus multidirectional balance training on muscle reaction time in subjects with chronic ankle instability. Muscle reaction time is measured on a trapdoor simulating an inversion sprain before and after a 6 week lasting balance training protocol.

ELIGIBILITY:
According to the consensus statement of the International Ankle Consortium

Inclusion Criteria:

* History of an ankle sprain
* Repetitive ankle sprains AND feelings of instability AND giving way
* Ankle functionality is documented (not as inclusion criteria)

Exclusion Criteria:

* Fracture
* Surgery
* equilibrium disorder

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
muscle reaction time | 6 weeks
  Muscle reaction of lower leg muscles is recorded during sudden simulated inversion sprain on a trap door

CONTACTS AND LOCATIONS:
Overall Officials: Roel De Ridder, Principal Investigator — University Ghent

IPD SHARING:
Plan to Share IPD: No